CLINICAL TRIAL: NCT06264453
Title: A Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel-designed, Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of KH001 in Patients with Dentin Hypersensitivity
Brief Title: A Study to Evaluate the Efficacy and Safety of KH001 in Patients with Dentin Hypersensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HysensBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KH-001-D201
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Dentin Hypersensitivity
Keywords: Dentin Sensitivity; Denin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): KH001 0.2mg/mL
  Interventions: Drug: KH001
- Group B (Experimental): KH001 0.4mg/mL
  Interventions: Drug: KH001
- Group C (Placebo Comparator): Water for Injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KH001 — topical applications of KH001
  Arms: Group A; Group B
Drug: Placebo — topical applications of Water for Injection
  Arms: Group C

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KH001 in patients with dentin hypersensitivity.

DETAILED DESCRIPTION:
This study is multicenter, double-blind, placebo-controlled, randomized, parallel-designed, phase 2 study to evaluate the efficacy and safety of KH001. The total duration of the study will be approximately 7 to 11 weeks. Clinical safety evaluations will include physical examinations, vital signs, clinical laboratory results, and Adverse Event monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 19 years old by the time of the screening visit
* Be in good general health as determined by the investigator
* Have at least 2 non-adjacent teeth and is diagnosed with hypersensitive

Exclusion Criteria:

* Is allergic to the active drug substance or other excipients used in the investigational product
* Has any history of alcohol or drug abuse
* Has received any treatment related to dentin hypersensitivity within 8 weeks prior to the screening visit
* Has active dental caries or history of dental caries

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Schiff sensitivity score | Baseline and Day 36
  Schiff sensitivity score 0-3 by air blast

SECONDARY OUTCOMES:
Change from baseline in a Schiff sensitivity score | Baseline, Day 8, 15, 22 and 43
  Schiff sensitivity score 0-3 by an evaporative air
Change from baseline in a Tactile threshold | Baseline, Day 8, 15, 22, 36 and 43
  Tactile threshold by yeaple probe
Change from baseline in Visual Analogue Scale | Baseline, Day 8, 15, 22, 36 and 43
  100mm Visual Analogue Scale

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung-Kyu Choi, D.D.S, Principal Investigator — Kyung Hee University Dentistry Hospital
Locations (1):
- Kyung Hee University Dental Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No